CLINICAL TRIAL: NCT06171412
Title: Glu-COACH: a Peer-mentoring Intervention to Reduce Disparities in Continuous Glucose Monitor (CGM) Use
Acronym: Glu-COACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000033606; 1R01DK134977-01 (NIH)
Record Dates: First submitted 2023-12-05; First posted 2023-12-14 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes
Keywords: continuous glucose monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glu-COACH (Experimental): The experimental group will receive ESOC plus peer-mentoring support from a peer of the same cultural identity (Glu-COACH) and access to a private social media group for all Black and Latinx teens to improve the initiation and maintenance of CGM (Dexcom)
  Interventions: Behavioral: Glu-COACH

INTERVENTIONS:
Behavioral: Glu-COACH — peer-mentoring support from a peer of the same cultural identity and access to a private social media group for all Black and Latinx teens

SUMMARY:
This is a study to develop and evaluate a peer mentoring intervention for Black and Latinx adolescents with type 1 diabetes to increase the initiation and maintenance of a continuous glucose monitoring (CGM) device. This device is a standard of care to improve diabetes management related to diet, exercise, and insulin. Use of CGM has been shown to improve health outcomes, but is not used by adolescents of color. Peer mentors may help improve usage.

DETAILED DESCRIPTION:
In Phase 1, investigators developed the intervention with a stakeholder advisory group. In Phase 2, investigators will conduct a small clinical trial to evaluate the intervention. Phase 1 is complete with the focus of this registration being Phase 2, the clinical trial.

All study procedures will be conducted remotely by ZOOM, including consent/assent, device and training, and peer mentor sessions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes, as determined clinically by the presence of ketosis or ketoacidosis at presentation and/or the presence of at least one diabetes-related auto-antibody
* Self-identification as Black and/or Latinx.
* Ability of participant to comprehend and communicate in written and spoken English, in order to complete surveys and participate in mentioning sessions and other interview (parents/caregivers do not need to have English fluency)
* Access to personal cellphone or tablet to participate in remote video sessions with the peer mentor
* using CGM <50% of the time over the last 3 months

Exclusion Criteria:

* Participants with a prior severe skin reaction to CGM sensor or adhesive.
* Current use of CGM
* Current or planned pregnancy
* Inability to comprehend or communicate in spoken/written English
* Subjects with other medical or mental health conditions that would, in the opinion of the investigators, interfere with the conduct of the study or present additional risk to the individual.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Mean hours per week CGM worn | 3 months and 6 months
  Mean hours per week of documented CGM wear. This will be documented through the CGM program. The primary analysis will be CGM use time at 6 months between the two groups.

SECONDARY OUTCOMES:
CGM Mean glucose | baseline, 3 months and 6 months
  The mean glucose in mg/dL
CGM Percentage time in range (70-180mg/dL) | baseline, 3 months and 6 months
  Percentage of time participants glucose values are in the target range of 70-180 mg/dL
Mean A1C concentration | baseline, 3 months and 6 months
  Mean A1C concentration
Number of Adverse diabetes-related events (diabetic ketoacidosis) | baseline, 3 months and 6 months
  Number of Yes/no responses via self report of diabetic ketoacidosis
Number of Adverse diabetes-related events (severe hypoglycemia) | baseline, 3 months and 6 months
  Number of Yes/no responses via self report of severe hypoglycemia
Mean score in Diabetes Distress using Problem Areas in Diabetes-Teen (PAID-T) survey | baseline, 3 months and 6 months
  PAID-T is a 26 item survey that measures of diabetes-specific distress for teenagers with type 1 diabetes. Items are rated on a 6-point Likert scale: 1-2, not a problem; 3-4, a moderate problem; or 5-6, a serious problem. Item scores are summed to form a total score (range 26-156), with higher scores indicating greater distress.
Mean score Diabetes self-efficacy using Diabetes Management Self-Efficacy scale (DMSES) | baseline, 3 months and 6 months
  Measures the diabetic patients confidence regarding diet, exercise and medical treatment. It is a 20 item survey. Responses are rated on a 5 point scale ranging from 1- ''can't do at all'' to 5- ''certain can do''. Item scores are summed to form a total score range 0-100 with higher scores indicating higher self-efficacy in performing diabetes self management activities.
Mean score Depressive symptoms using Patient Health Questionnaire-2 (PHQ-2) | baseline, 3 months and 6 months
  The PHQ-2 is a 2 item questionnaire used to assess the frequency of depressed mood. Item scores are summed with a total score ranging from 0 to 6 with higher scores indicating higher frequency of depressed moods.
Mean score Anxiety symptoms using General Anxiety Disorder-7 (GAD-7) | baseline, 3 months and 6 months
  General Anxiety Disorder- 7 (GAD-7) is a 7 item self report instrument that measures anxiety. Items are scored on a 4-point scale, ranging from "not at all (0)" to "nearly everyday (3)". Item scores are summed with a total score ranging from 0 to 21: 0-4 Minimal anxiety; 5-9 Mild anxiety; 10-14 Moderate anxiety; 15-21 Severe anxiety.
Mean score Family conflict using Diabetes Family Conflict Scale (DFCS) | baseline, 3 months and 6 months
  DFCS is a 19-item measure of diabetes management and the implications it has on the caregiver-child relationship. Items are scored on a 3-point Likert scale (1 = never argue, 2 = sometimes argue, and 3 = always argue). Item scores are summed with a total scale range of 19 to 57 with higher scores indicating a higher level of conflict.
Mean score Benefits and burdens of CGM use | baseline, 3 months and 6 months
  This survey consists of two sub-scales (one is benefits, one is burdens) with 8 items each. Each item scored Likert scale - Scored 1-5 Strongly Disagree to Agree. Items summed and divided by # of items. Mean score across participants. Each subscale range 1-5, with 5 indicating greater perceived benefits or burdens.
Mean Score Technology Attitudes | baseline, 3 months and 6 months
  5 items scored on a Likert scale, scored 1-5 (strongly disagree to agree). Items summed and divided by # of items. Mean score across participants. Score range 1-5, with 5 indicating more positive attitude about technology.
Mean score Glu-Coach satisfaction scale | 3 months and 6 months
  5 items scored on a Likert scale, scored 1-5 (not at all to extremely). Items summed and divided by # of items. Mean score across participants. Score range 1-5, with 5 indicating greater satisfaction.
Mean count Barriers to Device Use | 3 months and 6 months
  19 items with yes/no response. Mean number of barriers across participants. Higher value indicates more barriers.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Whittemore, PhD, APRN, FAAN, Principal Investigator — Yale School of Nursing; Stuart A Weinzimer, MD, Principal Investigator — Yale University
Locations (1):
- Yale Children's Diabetes Clinic, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data associated with the study, upon request for qualified academic investigators for non-commercial use. Meta-analysis data along with data content, format, and organization, will be available on request. Submitted data will comply with relevant data and terminology standards.
  De-identified data will be made available upon request by the study principal investigators, and that these data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA). Names and Institutions of persons either given or denied access to the data, and the bases for such decisions, will be summarized in the annual progress report.
  Data and secondary analysis of data will be maintained in a secure data-base on the Yale system.
Supporting Information: Study Protocol, SAP
Time Frame: After completion of the funded project period for the parent award and upon acceptance of the data for publication.
Access Criteria: Investigators agree to identify where the data will be available and how to access the data in any publications and presentations that the investigators author or co-author about these data, as well as acknowledge the funding source in any publications and presentations.